CLINICAL TRIAL: NCT03281967
Title: Clinical Survey of Minimally Invasive Ponto Surgical Technique (MIPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C63
Record Dates: First submitted 2017-08-31; First posted 2017-09-13 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bone Conduction Deafness; Unilateral Deafness; Middle Ear Deafness; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally Invasive Ponto Surgery (Other): Surgical method for installation of a bone anchored hearing system for hearing rehabilitation
  Interventions: Device: Minimally Invasive Ponto Surgery

INTERVENTIONS:
Device: Minimally Invasive Ponto Surgery — Minimally Invasive Ponto surgery is used for hearing rehabilitation using Ponto Wide Implant in patients indicated and counselled for Bone Anchored Hearing System.

SUMMARY:
The objective of the study is to compare the outcomes after a surgical procedure with minimally invasive Ponto surgery (MIPS, test group) and tissue preservation surgery (control) for placing Oticon Medical Ponto implants and abutments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patient indicated for an ear level bone anchored sound processor.
* Healthy bone quality to allow for 4mm implant insertion.

Exclusion Criteria:

* Intraoperative switch to an alternative surgical technique
* Patients undergoing re-implantation (on the side being included in the study)
* Previous participation in the C47 study.
* Inability to participate in follow-up.
* Psychiatric disease in the medical history.
* Mental disability.
* Presumed doubt, for any reason, that the patient will be able to show up on all follow-ups.
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.
* Patients with natural skin height of >12mm (as there will be additional skin reduction needed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Numbness (sensibility) around surgery area | 6 months post surgery
  The primary objective of the study is to investigate the difference in numbness around implant after MIPS procedure (test, this investigation) and a surgery with soft tissue preservation (control, from a previous study, C47) for implanting Oticon Medical implants and abutments.
  Two different sensibilities will be tested by means of a broken wooden cotton swab/bud (q-tip): gnostic (with cotton side) and vital (with broken, sharp wooden side) sensibility. The measurement locations will be standardized at specific positions from surgery location, and the same location (with respect to the surgery site) will be used for sensibility measurement for each patient visit. Both the area (diameter in cm) and the degree (scale form 0 (no complaints) to 10 (maximum complaints)) will be monitored. Additionally, patients' subjective sensibility judgment around surgery area on a scale of 0-10 will be recorded.

SECONDARY OUTCOMES:
Time needed for surgery | At surgery
  Compare the surgical time between test (this investigation) and control group (previous investigation, C47).
Unplanned visit | 36 months
  Investigate and compare the number of unplanned visits, unplanned surgical procedures and other treatments for the test (this investigation) and control group (previous investigation, C47).
Adverse Events | 36 months
  Investigate and compare the rate of adverse skin reactions using the Holgers Scale and the IPS scale.
Pain perception by patient | 36 months
  Investigate and compare patient perceived pain.
  For pain measurement, the patient is asked if pain around the implant is present. If it's present, duration is assessed (more or less than 6 weeks present). In addition, increase of pain is assessed during manipulation of the abutment (tightening of or tapping on the abutment). The patient is asked to score the perceived pain on a scale of 0-10; with 0 being no pain at all and 10 being the highest pain the patient had ever experienced.
Implant survivability | 36 months
  Investigate and compare implant survivability.
  Implant survivability is monitored by following upon patients and recording implant losses if and when they occur. The investigators do not expect multiple patients to have an implant loss. However, this may happen due to different reasons. The investigators would track the circumstances under which the implant loss occurred and the time between implant installation and loss.
Implant stability as measures by Implant stability quotient. | 36 months
  Investigate implant stability.
Surgical wound healing time | 36 months
  Investigate and compare healing time after surgery.
  Follow-up visits after surgery will assess the healing of wound. This will be a yes/no assessment to be answered by the attending physician. The investigators will also evaluate skin reactions using the Holgers Scoring Scheme and record any medications that were given to aid in skin healing.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by APHAB, GBI and GHSI questionnaires.
Aesthetic Assessment | 36 months
  Investigate and compare scar assessment by surgeon and patient (POSAS).

CONTACTS AND LOCATIONS:
Overall Officials: Myrthe Hol, MD, PhD, Principal Investigator — Radboud UMC, Department of Otorhinolaryngology. The Netherlands
Locations (1):
- University Medical Center St Radboud, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No